CLINICAL TRIAL: NCT06586125
Title: The Impact of Virtual Reality on Powered Mobility in Patients With Neuromotor Disabilities: a Feasibility Study
Brief Title: Virtual Reality Impact on Powered Mobility: a Feasibility Study
Acronym: VR-PMP
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: 002.2022.ISNB.NeuroRehab.MRI
Record Dates: First submitted 2024-06-28; First posted 2024-09-19 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy Infantile; Neuromuscular Diseases in Children
Keywords: Cerebral palsy; Neuromuscular diseases; Powered mobility; Virtual reality; Pediatric rehabilitation; Brain-computer interface
MeSH Terms: conditions — Cerebral Palsy; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VR - based training: Five children and adolescents with cerebral palsy and/or neuromuscular disease and five children and adolescents with cerebral palsy and/or neuromuscular disease with difficulties to control the VR joysticks
  Interventions: Other: Powered Mobility Training

INTERVENTIONS:
Other: Powered Mobility Training — The study procedure aims to observe the partecipants' behaviour while using the Virtual Reality - Power Mobility Program (VR-PMP) simulator applied during Power Mobility Training in clinical practice for 15 sessions. Participants use either semi-immersive mode (laptop screen with VR-PMP simulator) or immersive mode (head-mounted display with VR-PMP simulator). Five out of ten children unable to use conventional VR controllers or alternative access technologies available on the market, use brain-computer interface (BCI) developed specifically for these children to control the VR-PMP simulator.
  Other Names: Virtual Reality - based powered mobility training

SUMMARY:
This study explores the potential of Virtual Reality (VR) technology to enhance powered wheelchair (PW) training for children diagnosed with Cerebral Palsy (CP) and neuromuscular diseases (NMDs). The primary objective is to improve mobility and independence by employing immersive VR games and simulations within a powered mobility program (PMP) framework. The research involve testing a VR-powered mobility program (VR-PMP) simulator, which integrates 3D gaming tailored with PMP tasks accessible via laptops or VR headsets. Specifically designed for children with severe movement limitations, the study incorporates Brain-Computer Interfaces (BCIs), enabling interaction within the VR environment without conventional controllers. The study aims to evaluate whether these innovative VR tools can facilitate safer and independent wheelchair navigation for these children.

DETAILED DESCRIPTION:
Children diagnosed with Cerebral Palsy (CP) and neuromuscular diseases (NMDs) often face significant challenges in achieving independent mobility due to motor impairments. Powered mobility is a viable option, but it requires extensive training to ensure safe driving conditions. Typically, wheelchair training is conducted with therapists at the hospital, incurring considerable costs for the national health system. Additionally, 10-40% of people are unable to use a power wheelchair due to sensory, motor, and neurocognitive impairments. These individuals are deemed unable to drive safely and are often forced to use manual wheelchairs or rely on caregivers for support. Driving skills and appropriate aids for independent mobility are established based on the Powered Mobility Program (PMP). However, to date, no clinically validated tools exist to support user training in fulfilling the PMP requirements.

Virtual reality (VR) offers a portable solution for safe training at home. However, current VR simulators have not been developed to assess users' driving skills, and they typically allow control via joysticks or hand trackers, which are unusable for individuals with severe upper limb motor impairments. In this context, brain-computer interfaces (BCIs) represent a potential innovative control interface.

Integrating VR into powered wheelchair (PW) training introduces new possibilities for enhancing rehabilitation programs by offering engaging and personalized experiences tailored to the unique needs of children with CP and NMDs. The VR Powered Mobility Program (VR-PMP), which integrates 3D gaming tailored to PMP tasks accessible via laptops or VR headsets, aims to harness the potential of VR to enhance PW training. VR-PMP seeks to facilitate motor learning through repetitive practice in realistic and engaging contexts.

The primary objective of this study is to assess the feasibility of using immersive and semi-immersive VR for powered mobility (PM) training and to determine the impact of VR technologies on PW driving skills in children with CP and NMDs, including those with severe upper limb motor impairments.

The secondary aims are:

To assess the impact of VR: evaluating the use of VR on the level of assistance, supervision, and autonomy in PW driving, measured through the overall PMP score, comparing PMP scores obtained before and after VR training to determine improvements in PW driving skills.

To correlate physiological signals collected during VR-PMP sessions with motion sickness and workload assessments to understand stress levels and engagement.

To investigate the usability and satisfaction with the VR PMP system through questionnaires and scales, focusing on the feasibility of home training sessions for driving practice.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age between 6 and 20 years
* Clinical diagnosis: Central motor disability with Gross Motor Function Classification Scale (GMFCS) levels 3-4-5
* Owner of a powered wheelchair or a manual wheelchair with an electric propulsion system
* Powered Mobility Program (PMP) score > 0 in basic skills
* Signed informed consent

Exclusion Criteria:

* Participants who do not tolerate the use of immersive VR (e.g., development of motion sickness-related symptoms)
* Severe cognitive impairments

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will enroll up to ten pediatric participants diagnosed with cerebral palsy (CP) or neuromuscular diseases (NMDs) who require powered wheelchair for their mobility.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of dropout participants unable to use the VR-PMP simulator | from Tprel (day 1) to T13 (day 41)
  This outcome assesses the capability of using the VR-PMP (Virtual Reality-Powered Mobility Program) simulator by observing dropout rates, from 0 participant to 10 participants due to technology issues (e.g., equipment usability, motion sickness), as well as satisfaction levels with VR (Virtual Reality) hardware and software.

SECONDARY OUTCOMES:
PMP (Powered Mobility Program) score | T0 (day 2), T1 (day 3), T6 (day 25), T12 (day 40), T13 (day 41)
  The Powered Mobility Program (PMP) score assesses assistance, supervision, and autonomy in driving powered wheelchairs through 34 tasks. These tasks are categorized into basic skills, structured environment driving, and unstructured environment driving domains. Each task is scored from 0 (task not attempted) to 5 (age-appropriate supervision), with a maximum total score of 170 points. The total score is calculated by summing individual item scores and dividing by the number of completed tasks.
QUEST-2 (Quebec User Evaluation of Satisfaction with Assistive Technology) questionnaire score | T0 (day 2), T13 (day41)
  The QUEST 2.0 questionnaire score is an outcome measurement that evaluates user's satisfaction with their assistive device. It is used to document the real-life benefits of assistive devices and justify their necessity. It comprises 12 items divided into two parts: Device (8 items) and Services (4 items). Each item is rated on a 5-point scale from 1 ("not satisfied at all") to 5 ("very satisfied"). The total score is the sum of valid item scores divided by the number of valid items.
MSAQ (Motion Sickness Assessment Questionnaire) score | T1 (day 3), T6 (day 25), T12 (day 40)
  The MSAQ questionnaire assesses motion sickness. It consists of 16 questions divided into four subcategories: Gastrointestinal (G), Central (C), Peripheral (P), and Sopite-related (S). Responses are scored on a scale from 1 to 9 points. Each subcategory is scored individually, contributing to a total score ranging from 11 to 144 points. The overall motion sickness score is calculated as the percentage of total points scored: (sum of all item points / 144) × 100. Subscale scores are calculated similarly as percentages within each factor: (sum of gastrointestinal items / 36) × 100; (sum of central items / 45) × 100; (sum of peripheral items / 27) × 100; (sum of sopite items / 36) × 100.
IPQ (iGroupPresence Questionnaire) score | T1 (day 3), T6 (day 25), T12 (day 40)
  The IPQ questionnaire assesses sense of presence (SOP - level of immersion in VR) of a VR user. The IPQ consists of 14 items divided into four subcategories: spatial presence, involvement, perceived realism level, and a "sense of being present." All items are rated on a seven-point scale (0-6), with a higher score indicating greater SOP. The total score is obtained by summing the scores of individual items (from 0 to 84 points).
NASA-TLX (NASA Task Load Index) score | T0 (day 2), T1 (day 3), T6 (day 25), T12 (day 40), T13 (day 41)
  The NASA-TLX questionnaire score (National Aeronautics and Space Administration Task Load Index) measures physical and mental workload using six items related to mental load, physical activity, speed of performance, performance, effort, and frustration. Each item is accompanied by a 12 cm line scale divided into 20 equal intervals, anchored by binary descriptors (e.g., low/high), delimited by 21 vertical markers, and then converted to a scale from 0 to 100 points. To calculate the score for each scale, the number of lines marked by a participant is counted, 1 is subtracted, and the result is multiplied by 5. Weights from 0-5 will be assigned to the 15 subscale comparisons, which will be multiplied by the corresponding subscale score. The total score (from 0 to 100 points) is estimated by summing the weighted scores and dividing by 15.
mNASA-TLX (modified NASA Task Load Index) score | T2 (day 6), T3 (day 12), T4 (day 18), T5 (day 24), T7 (day 26), T8 (day 30), T9 (day 33), T10 (36), T11 (39)
  Participants will be asked to fill out a modified version of the NASA-TLX (mNASA-TLX), using the same questions but with a different scale ranging from 1 (low) to 5 (high). The scores will be then converted using the 0-100 points scale, as for the NASA-TLX.
GDQ (Game Design Questionnaire) score | T1 (day 3), T6 (day 25), T12 (day 40)
  The GDQ is a questionnaire to evaluate the user's satisfaction of the VR-PMP simulator. It assesses the usability of the graphical interface and user preferences (measured on a scale from 1 to 9 points) regarding colors, game animation, and avatars used. The total score is estimated by averaging the items.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Cersosimo, Dr., Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna
Locations (1):
- IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Background] Mercuri E, Muntoni F. Muscular dystrophies. Lancet. 2013 Mar 9;381(9869):845-60. doi: 10.1016/S0140-6736(12)61897-2. PMID 23465426
- [Background] Jones MA, McEwen IR, Neas BR. Effects of power wheelchairs on the development and function of young children with severe motor impairments. Pediatr Phys Ther. 2012 Summer;24(2):131-40; discussion 140. doi: 10.1097/PEP.0b013e31824c5fdc. PMID 22466379
- [Background] Rosen L, Plummer T, Sabet A, Lange ML, Livingstone R. RESNA position on the application of power mobility devices for pediatric users. Assist Technol. 2023 Jan 2;35(1):14-22. doi: 10.1080/10400435.2017.1415575. Epub 2018 Mar 26. PMID 29232181
- [Background] Bottos M, Bolcati C, Sciuto L, Ruggeri C, Feliciangeli A. Powered wheelchairs and independence in young children with tetraplegia. Dev Med Child Neurol. 2001 Nov;43(11):769-77. doi: 10.1017/s0012162201001402. PMID 11730152
- [Background] Bray N, Kolehmainen N, McAnuff J, Tanner L, Tuersley L, Beyer F, Grayston A, Wilson D, Edwards RT, Noyes J, Craig D. Powered mobility interventions for very young children with mobility limitations to aid participation and positive development: the EMPoWER evidence synthesis. Health Technol Assess. 2020 Oct;24(50):1-194. doi: 10.3310/hta24500. PMID 33078704
- [Background] Livingstone R, Field D. Systematic review of power mobility outcomes for infants, children and adolescents with mobility limitations. Clin Rehabil. 2014 Oct;28(10):954-64. doi: 10.1177/0269215514531262. Epub 2014 Apr 24. PMID 24764156
- [Background] Kirby RL, Dupuis DJ, Macphee AH, Coolen AL, Smith C, Best KL, Newton AM, Mountain AD, Macleod DA, Bonaparte JP. The wheelchair skills test (version 2.4): measurement properties. Arch Phys Med Rehabil. 2004 May;85(5):794-804. doi: 10.1016/j.apmr.2003.07.007. PMID 15129405
- [Background] Gefen N, Weiss PL, Rigbi A, Rosenberg L. Lessons learned from a pediatric powered mobility lending program. Disabil Rehabil Assist Technol. 2024 Aug;19(6):2250-2259. doi: 10.1080/17483107.2023.2276232. Epub 2023 Oct 28. PMID 37897432
- [Background] Field DA, Livingstone RW. Power mobility skill progression for children and adolescents: a systematic review of measures and their clinical application. Dev Med Child Neurol. 2018 Oct;60(10):997-1011. doi: 10.1111/dmcn.13709. Epub 2018 Mar 14. PMID 29542110
- [Background] Fraudet B, Leblong E, Piette P, Nicolas B, Gouranton V, Babel M, Devigne L, Pasteau F, Gallien P. Evaluation of power wheelchair driving performance in simulator compared to driving in real-life situations: the SIMADAPT (simulator ADAPT) project-a pilot study. J Neuroeng Rehabil. 2024 Apr 23;21(1):60. doi: 10.1186/s12984-024-01354-5. PMID 38654367
- [Background] Faure C, Routhier F, Lettre J, Choukou MA, Archambault PS. Effectiveness of the miWe Simulator Training on Powered Wheelchair-driving Skills: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 Sep;104(9):1371-1377. doi: 10.1016/j.apmr.2023.04.022. Epub 2023 May 19. PMID 37209934
- [Background] Furumasu J, Guerette P, Tefft D. Relevance of the Pediatric Powered Wheelchair Screening Test for children with cerebral palsy. Dev Med Child Neurol. 2004 Jul;46(7):468-74. doi: 10.1017/s0012162204000775. PMID 15230460
- [Background] Gefen N, Archambault PS, Rigbi A, Weiss PL. Pediatric powered mobility training: powered wheelchair versus simulator-based practice. Assist Technol. 2023 Sep 3;35(5):389-398. doi: 10.1080/10400435.2022.2084183. Epub 2022 Jun 23. PMID 35737961
- [Background] Gefen N, Rigbi A, Weiss PLT. Reliability and validity of pediatric powered mobility outcome measures. Disabil Rehabil Assist Technol. 2022 Nov;17(8):882-887. doi: 10.1080/17483107.2020.1819449. Epub 2020 Sep 12. PMID 32924663
- [Background] Gefen N, Rigbi A, Archambault PS, Weiss PL. Comparing children's driving abilities in physical and virtual environments. Disabil Rehabil Assist Technol. 2021 Aug;16(6):653-660. doi: 10.1080/17483107.2019.1693644. Epub 2019 Dec 5. PMID 31805790
- [Background] Gefen N, Rigbi A, Weiss PL. Predictive model of proficiency in powered mobility of children and young adults with motor impairments. Dev Med Child Neurol. 2019 Dec;61(12):1416-1422. doi: 10.1111/dmcn.14264. Epub 2019 May 21. PMID 31115048
- [Background] Gefen N, Rosenberg L. Development of a new tool: progression of paediatric powered mobility- 3PM. Disabil Rehabil Assist Technol. 2024 Feb;19(2):465-473. doi: 10.1080/17483107.2022.2099020. Epub 2022 Jul 14. PMID 35833624
- [Background] Demers L, Weiss-Lambrou R, Ska B. Item analysis of the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST). Assist Technol. 2000;12(2):96-105. doi: 10.1080/10400435.2000.10132015. PMID 11508406
- [Background] Gianaros PJ, Muth ER, Mordkoff JT, Levine ME, Stern RM. A questionnaire for the assessment of the multiple dimensions of motion sickness. Aviat Space Environ Med. 2001 Feb;72(2):115-9. PMID 11211039
- [Background] Salimi Z, Ferguson-Pell MW. Motion sickness and sense of presence in a virtual reality environment developed for manual wheelchair users, with three different approaches. PLoS One. 2021 Aug 19;16(8):e0255898. doi: 10.1371/journal.pone.0255898. eCollection 2021. PMID 34411151
- [Background] Laurie-Rose C, Frey M, Ennis A, Zamary A. Measuring perceived mental workload in children. Am J Psychol. 2014 Spring;127(1):107-25. doi: 10.5406/amerjpsyc.127.1.0107. PMID 24720100